CLINICAL TRIAL: NCT05508165
Title: IRB: #12530 Prospective, Randomized Study to Assess Clinical Outcomes and Patient Satisfaction of Virtual vs. In-Person Workup and Treatment of Lower Urinary Tract Symptoms
Brief Title: Patient Satisfaction of Virtual vs In-Person Workup and Treatment of Lower Urinary Tract Symptoms.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Marcelino Rivera, Assistant Professor, IU Department of Urology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IndianaU 12530
Record Dates: First submitted 2022-05-02; First posted 2022-08-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Urologic Diseases
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cohort 1a: in-person clinical assessment of LUTS/BPH (No Intervention): COHORT 1a: Subjects randomized to undergo in-person initial clinical workup of Lower Urinary Tract Symptoms (LUTS) / Benign Prostatic Hyperplasia (BPH) and in-person clinical follow-up after 3 months of clinical intervention. In-person clinical workup at both the initial and Month 3 follow-up timepoint includes International Prostate Symptom Score (IPSS), and standard of care uroflowmetry, post void residual (PVR), and urinalysis (UA) assessments.
- Cohort 1b: virtual (telehealth) clinical assessment of LUTS/BPH (Experimental): COHORT 1b: Subjects randomized to undergo virtual initial clinical workup of Lower Urinary Tract Symptoms (LUTS) / Benign Prostatic Hyperplasia (BPH) and virtual clinical follow-up after 3 months of clinical intervention. Virtual clinical workup at both the initial and Month 3 follow-up timepoint includes at home completion of International Prostate Symptom Score (IPSS), at home uroflowmetry assessment through use of the Stream Dx device, at home assessment of post void residual (PVR) through use of the DFree device, and at home urinalysis (UA) through use of the TestCard device.
  Interventions: Device: Stream Dx; Device: DFree; Device: TestCard
- Cohort 2: Validation Cohort (Other): COHORT 2: Non-randomized subjects who will attend a single, clinically scheduled, in-person follow-up appointment to directly compare the standard of care assessments/devices to the experimental assessments/devices. Prior to the in-person appointment, patients will complete at home uroflowmetry assessment through use of the Stream Dx device. At the in-person appointment, the clinic staff will perform standard of care uroflowmetry, post void residual (PVR), and urinalysis (UA). At this visit, clinic staff will also obtain PVR measurements through use of the DFree device and urinalysis through the TestCard device.
  Interventions: Device: Stream Dx; Device: DFree; Device: TestCard

INTERVENTIONS:
Device: Stream Dx — home uroflowmetry device
  Arms: Cohort 1b: virtual (telehealth) clinical assessment of LUTS/BPH; Cohort 2: Validation Cohort
Device: DFree — at home wearable bladder scanner
  Arms: Cohort 1b: virtual (telehealth) clinical assessment of LUTS/BPH; Cohort 2: Validation Cohort
Device: TestCard — mobile urinalysis reader
  Arms: Cohort 1b: virtual (telehealth) clinical assessment of LUTS/BPH; Cohort 2: Validation Cohort

SUMMARY:
This study is being done to compare usefulness of data collected in uroflowmetry, a test that measures the amount of urine released from the body, at home versus in the doctor's office. Additionally, investigators are assessing patient satisfaction when completing a virtual visit for lower urinary tract symptoms (LUTS), related to prostatic enlargement, compared to an in person visit.

The three devices being investigated have not been used in the home setting to make urinary measurements as is typically done in clinic. The goal is to test the effectiveness and accuracy of these devices compared to our standard clinical practices and demonstrate their ability to provide useful information in the home setting.

DETAILED DESCRIPTION:
This study is being done to improve the availability of telehealth urology visits. In this study, investigators will compare the usefulness of data collected by three home devices to understand the amount of urine released from the body, how empty the bladder gets after urinating, and if there is an infection present in the bladder. These will be compared to being at home versus in the doctor's office. Additionally, the study will determine how satisfied patients are when completing a virtual visit for lower urinary tract symptoms (LUTS), related to prostatic enlargement, compared to an in-person visit. The three devices being investigated have not been used in the home setting to make urinary measurements as is typically done in clinic. The goal is to test the effectiveness and accuracy of these devices compared to standard clinical practices and demonstrate the ability of these devices to provide useful information in the home setting. The study involves two cohorts. Cohort 1 are new patients who will be randomized to either telehealth visits or in office visits. If randomized to the telehealth group, the patients will use various devices to perform a standard workup at home. If randomized to the clinic visit, similar tests will be performed in the office. Cohort 2 are existing patients who will use one of the devices at home, but will also complete similar in-office tests in order to compare device accuracy.

Screening will be performed prior to patient's first scheduled visit based on chief complaints of urinary retention, BPH, or LUTS. Patients will be initially identified by study personnel or qualified research coordinator when the patient is identified to have qualifying issues through reviewing medical records of patients. Patient will be contacted by phone by the study personnel. If the patients are interested, the patients will be screened for inclusion criteria.

ELIGIBILITY:
Inclusion Criteria

* ≥18 years of age
* New patient referral for urinary retention, BPH, or LUTS (Cohort 1)
* Established patient for urinary retention, BPH, or LUTS (Cohort 2)
* Male

Exclusion Criteria

* <18 years of age
* Inability to provide informed consent
* Visually or hearing impaired
* Concomitant condition requiring in-person exam or evaluation
* History of allergic reaction or issues with ultrasound gel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) Baseline | Baseline
  The IPSS assesses prostate related symptoms and their frequency of occurrence through seven questions, scored on a 6 point scale, from 0 (not at all) to 5 (always). Total symptom-related scores range from 1-7 (mild), 8-19 (moderate), and 20-35 (severe). The IPSS also assess quality of life due to urinary symptoms with a single question, scored on a 7 point scale (0 = delighted; 6 = terrible).
  The IPSS will be administered at the initial visit (baseline) for Cohorts 1a and 1b. Baseline scores will be compared between the two groups to evaluate for equivalency.
International Prostate Symptom Score (IPSS) Change | 3 months
  The IPSS assesses prostate related symptoms and their frequency of occurrence through seven questions, scored on a 6 point scale, from 0 (not at all) to 5 (always). Total symptom-related scores range from 1-7 (mild), 8-19 (moderate), and 20-35 (severe). The IPSS also assess quality of life due to urinary symptoms with a single question, scored on a 7 point scale (0 = delighted; 6 = terrible).
  The IPSS will be administered at the initial visit (baseline) and Month 3 for Cohorts 1a and 1b. The amount of IPSS score reduction at the time of 3 month follow up will be compared between both groups to evaluate for equivalency.
Uroflowmetry Baseline | Baseline
  Uroflowmetry measures the flow of urine as milliliters (ml) of urine passed per second(s). Typical scores range between 5 and 20 ml/s, with a lower score indicating possible obstruction, enlarged prostate or weak bladder and a higher score indicating good flow.
  Cohort 1a will undergo in-person uroflowmetry per standard clinical assessment at Baseline. Standard clinical assessment includes measurement of a single void during the in-person clinic visit by urinating once into the uroflowmetry device (a urinal with calibrated sensors to measure flow).
  Cohort 1b will undergo uroflowmetry through at-home use of the Stream Dx device (also a urinal with calibrated sensors to measure flow), which includes measuring all voids performed at home during a 5 day period prior to Baseline (initial virtual visit).
  Baseline uroflowmetry assessment results for Cohorts 1a and 1b will be evaluated for equivalency.
Uroflowmetry Change | 3 months
  Uroflowmetry measures the flow of urine as milliliters (ml) of urine passed per second(s). Typical scores range between 5 and 20 ml/s, with a lower score indicating possible obstruction, enlarged prostate or weak bladder and a higher score indicating good flow.
  Cohort 1a will undergo in-person uroflowmetry per standard clinical assessment at Baseline and Month 3. Standard clinical assessment includes measurement of a single void during the in-person clinic visit by urinating once into the uroflowmetry device.
  Cohort 1b will undergo uroflowmetry through at-home use of the Stream Dx device (also a urinal with calibrated sensors to measure flow), which includes measuring all voids performed at home during a 5 day period prior to Baseline (initial virtual visit) and again during a 5 day period prior to the Month 3 follow up visit.
  Increase in average flow at 3 months on uroflowmetry for Cohorts 1a and 1b will be evaluated for equivalency.
Post Void Residual (PVR) Baseline | Baseline
  Post Void Residual is the amount of urine remaining in the bladder after voiding. Typical scores range between 0 and 150 mL, with a higher score indicating incomplete bladder emptying.
  Cohort 1a will undergo in-person PVR assessment per clinical standards once at Baseline. This includes measurement of a single PVR volume during the clinical in-person visit using a calibrated ultrasound based bladder scanner that is placed on the patient's lower abdomen for 5 seconds.
  Cohort 1b will undergo PVR assessment through at-home use of the DFree device, a wearable bladder scanner. Participants will wear this device for an entire day during which will collect PVR measurements after each void during that period prior to the Baseline visit (initial virtual visit).
  PVR results for Cohorts 1a and 1b at baseline will be evaluated for equivalency.
Post Void Residual (PVR) Change | Baseline and 3 months
  Post Void Residual is the amount of urine remaining in the bladder after voiding. Typical scores range between 0 and 150 mL, with a higher score indicating incomplete bladder emptying.
  Cohort 1a will undergo in-person PVR assessment per clinical standards once at Baseline and Month 3 . This includes measurement of a single PVR volume during the clinical in-person visit using a calibrated ultrasound based bladder scanner that is placed on the patient's lower abdomen for 5 seconds.
  Cohort 1b will undergo PVR assessment through at-home use of the DFree device, a wearable bladder scanner. Participants will wear this device for an entire day during which will collect PVR measurements after each void during that period prior to the Baseline (initial virtual visit) and Month 3 virtual visit.
  Reduction in PVR between each group at the time of 3 month follow up will be evaluated for equivalency.
Urinalysis (UA) Baseline | Baseline
  Urinalysis (UA) the urine for infection (UTI) or diabetes. Recorded outcomes will be possible UTI (any positive leukocyte esterase, nitrites, or blood) and possible diabetes (any positive glucose, ketones, or proteins).
  Cohort 1a will undergo a UA assessment per standard clinical assessment once at the initial visit (baseline). This includes dipping a urine sample with a test strip which is read by a machine during the clinic in-person visit.
  Cohort 1b will undergo a UA assessment per standard clinical assessment once at the first virtual visit (baseline). Using the Testcard phone app, the patient will collect a urine sample at home, and dip a test strip into the urine which is then analyzed by the mobile app.
  UA results for Cohorts 1a and 1b will be evaluated for equivalency between the two groups at baseline. Any positive results (UTI or diabetes) will undergo confirmatory lab testing per standard of care.
Urinalysis (UA) 3 Months | 3 months
  Urinalysis (UA) the urine for infection (UTI) or diabetes. Recorded outcomes will be possible UTI (any positive leukocyte esterase, nitrites, or blood) and possible diabetes (any positive glucose, ketones, or proteins).
  Cohort 1a will undergo a UA assessment per standard clinical assessment once at Month 3 follow up. This includes dipping a urine sample with a test strip which is read by a machine during the clinic in-person visit.
  Cohort 1b will undergo a UA assessment per standard clinical assessment once at the Month 3 follow up. Using the Testcard phone app, the patient will collect a urine sample at home, and dip a test strip into the urine which is then analyzed by the mobile app.
  UA results for Cohorts 1a and 1b will be evaluated for equivalency between the two groups at 3 month follow up. Any positive results (UTI or diabetes) will undergo confirmatory lab testing per standard of care.

SECONDARY OUTCOMES:
Urology Satisfaction with Outpatient Service (SWOPS) baseline | Baseline
  Patient satisfaction in Cohorts 1a and 1b will be measured with the validated Satisfaction with Outpatient Service (SWOPS) questionnaire following their initial visit (baseline). The questionnaire assesses the patient's satisfaction with their visit across 13 topics. The investigators will test non-inferiority in SWOPS scores between patients in the virtual group and in-clinic group at the initial visit.
  There is no defined scale or score that would suggest a better or worse outcome, rather the percent response of "Yes, definitely", "Yes, to some extent", and "No" to each of the 13 questions will be compared between the two groups for equivalency and thus the non-inferiority statistical approach was chosen.
Urology Satisfaction with Outpatient Service (SWOPS) 3 months | 3 months
  Patient satisfaction in Cohorts 1a and 1b will be measured with the validated Satisfaction with Outpatient Service (SWOPS) questionnaire following their 3 month follow up. The questionnaire assesses the patient's satisfaction with their visit across 13 topics. The investigators will test non-inferiority in SWOPS scores between patients in the virtual group and in-clinic group at the initial visit.
  There is no defined scale or score that would suggest a better or worse outcome, rather the percent response of "Yes, definitely", "Yes, to some extent", and "No" to each of the 13 questions will be compared between the two groups for equivalency and thus the non-inferiority statistical approach was chosen.

OTHER OUTCOMES:
Stream Dx Device Validation | Baseline
  Cohort 2 will be asked to complete at home uroflowmetry assessment through use of the Stream Dx device for 5 days, starting 3 weeks prior to a single in-person clinical appointment to establish the baseline for that patient. During the in-person clinical appointment, Cohort 2 will also undergo standard uroflowmetry measurement by urinating once into the uroflowmetry device in the clinic (a urinal with calibrated sensors to measure flow). The baseline Stream Dx results including average and maximum flow rate in mL/s and volume voided in mL will be compared to those obtained by the in-person clinic performed uroflowmetry.
DFree Device Validation | Baseline
  Once at a single in-person clinical appointment, Cohort 2 will be asked to undergo a baseline assessment of post-void residual by both the standard clinic bladder scanner and the DFree device. Clinical staff will perform both the bladder scanner and DFree measurements. Baseline results between the assessment methods will be compared.
TestCard Device Validation | Baseline
  Once at a single in-person clinical appointment, Cohort 2 will be asked to undergo a baseline urinalysis assessment by both standard in clinic urinalysis dip stick and through the TestCard mobile app analysis. Clinical staff will perform both the standard and TestCard assessment on a single urine sample. Baseline results between the assessment methods will be compared. Recorded outcomes will be possible UTI (any positive leukocyte esterase, nitrites, or blood) and possible diabetes (any positive glucose, ketones, or proteins) and any positive results (UTI or diabetes) will undergo confirmatory lab testing per standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelino Rivera, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No